CLINICAL TRIAL: NCT01416246
Title: Pilot Trial of Fractionated Stem Cell Infusions in Myeloma Patients Undergoing Autologous Stem Cell Transplant
Brief Title: Fractionated Stem Cell Infusions in Myeloma Patients Undergoing Autologous Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-105
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma
Keywords: Stem cell Infusions; Autologous Stem Cell Transplant; 11-105
MeSH Terms: conditions — Multiple Myeloma | interventions — Erythrocyte Count; Platelet Transfusion; Therapeutics

ARMS (1):
- Fractionated Stem Cell Infusions (Experimental): A single arm, open-label, single institution pilot trial is planned. Patients with chemosensitive MM and at least 7 x 10^6 CD34+ stem cells/kg (+/- 0.5 x 10^6 CD34+ stem cells/kg)available for use will be enrolled following initial induction or salvage therapy.
  Interventions: Procedure: Fractionated Stem Cell Infusions

INTERVENTIONS:
Procedure: Fractionated Stem Cell Infusions — Following enrollment patients will be treated with melphalan intravenously (IV) through a central venous catheter (CVC) over 30 minutes at 200mg/m2 or 140mg/m2 (if creatinine clearance is < or = to 50 and/or age > 70 years) on day -2. Following 24 hours of rest, the first dose of CD34+ stem cell will be administered on day 0 (2.5-5 x 106 CD 34+ stem cells/kg)+/- 0.5 x 106 CD34+ stem cells/kg), followed by 3 additional doses of CD 34+ stem cells (1.5-2.5 x 106 CD 34+ stem cells/kg)+/- 0.5 x 106 CD34+ stem cells/kg) on days +2, +4, and +6. Pegfilgrastim 6μg will be administered on day +1. Filgrastim 5μg/kg will be 12-24 hours after the 2nd-4th stem cell infusions. There will be a +/- 1 day window for the Day +2, +4, and +6 infusions to accommodate infusions that occur over the weekend or on holidays.
  Other Names: Patients will receive standard supportive care measures (including; antimicrobial prophylaxis, red blood cell and platelet transfusions and; treatment for neutropenic fever) as per institutional practices. Neutrophil; engraftment is defined as absolute neutrophil count (ANC) > or = to 500 x 10^6/L for 2; consecutive days.

SUMMARY:
Multiple myeloma is difficult to treat with only anti-cancer medicine (called chemotherapy) or radiation alone. Sometimes higher doses of chemotherapy are used but when used can also lower blood counts. Using own cells (special cells called stem cells) to help increase the blood counts after high doses of chemotherapy is called autologous stem cell transplantation (ASCT).

Using own stem cells to restore blood counts and other advances in supportive measures (antibiotics and growth factors that increase blood counts) has improved the safety of ASCT. However, blood counts still decrease for a period of days after high doses of chemotherapy. During that time, patients are at greater risk for infections. Studies have shown that the faster the blood counts recover after ASCT, the less at risk there is for developing unwanted side effects after ASCT.

Typically during an ASCT, a patient's stem cells are given back to them all at once on a single day. In this study, the investigators plan to see what happens when smaller amounts of own stem cells are given back to the patient over multiple days. The investigators want to find out what effects good and/or bad this will have on the patient and there multiple myeloma. Some studies have shown that giving back stem cells over a period of days helps to increase bone marrow activity and decrease the time it takes for blood counts to recover after ASCT. It is our hope that this new approach may lower a patient's risk of side effects and infections, decrease the number of blood transfusions that a patient needs during this process, reduce the time a patient has to spend in the hospital, and lower overall treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and < than or = to 75
* Histologic and serologic findings, reviewed at MSKCC, confirming the diagnosis of multiple myeloma. Standard diagnostic criteria for multiple myeloma will be used, as per the International Myeloma Foundation consensus guidelines (Durie et al, 2003) .
* Patients must have symptomatic multiple myeloma who have responded to prior induction or salvage chemotherapy (i.e. chemosensitive disease):

  * Patients who are receiving high-dose melphalan and ASCT as part of their initial therapy require at least minor response to their last line of therapy to document chemosensitive disease (Anderson et al. 2008)
  * Patients who are receiving high-dose melphalan and ASCT as part of salvage therapy require at least a minor response to their last line of therapy to document chemosensitive disease (Anderson et al. 2008).
  * There is no limit on the number of prior regimens received by the patient.

    * Patients must have at least 7 x 10^6 (+/- 0.5 x 10^6) CD34+ stem cells/kg frozen if he/she is being treated as part of a salvage (second) transplant strategy; patients must have 10 x 10^6 (+/- 0.5 x 10^6) CD34+ stem cells/kg frozen if ASCT is being performed as part of initial therapy.
    * Adequate organ function is required, defined as follows:
  * Serum bilirubin ≤ 2.0 mg/dl
  * AST, ALT and alkaline phosphatase < 3 times the upper limit of laboratory normal
  * Creatinine clearance > or = to 40 ml/min (24 hour urine collection or calculated*)

    *To be calculated by the Cockroft-Gault method: (140-Age) x Mass (kg) x [0.85 if female] (72 x Creatinine (mg/dL)
  * LVEF > or = to 45% by MUGA or rest ECHO
  * Diffusing capacity > or = to 45% (adjusted for hemoglobin) predicted by pulmonary function testing
* Performance status KPS > or = to 70%.

Exclusion Criteria:

* Unstable angina or myocardial infarction within 4 months of initiating therapy on trial, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* Pregnant or lactating females
* Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Contraindication to melphalan or any of the required supportive treatments, including hypersensitivity to G-CSF or pegfilgrastim
* Any other medical condition or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
engraftment kinetics | 2 years
  as measured by duration of neutropenia in patients with MM undergoing high-dose melphalan followed by fractionated CD34+ stem cell infusions.

SECONDARY OUTCOMES:
safety and toxicity profile | 2 years
  of high-dose melphalan therapy followed by multiple doses of CD34+ stem cell rescue in patients with MM. Whenever possible, the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 should be used to describe the event and for assessing the severity of AEs.
neutrophil and platelet recovery rates. | 2 years
  Duration of neutropenia will be defined as the number of days ANC< 500x106/L. Time until platelet recovery (defined as platelets>=30x109/L), the number of units of red blood cells and platelets.
incidence of infection | 3 months post-SCT
  The incidence of infection by three months after re-infusion will be calculated.
red cell and platelet transfusion requirements | 2 years
  will be evaluated using the Spearman rank correlation coefficient
duration of hospital admission | 2 years
  length of hospital stay in days will be summarized using descriptive statistics.
To assess symptom burden | 2 years
  using the MSK Modified M.D. Anderson Symptom Inventory (MDASI).
Multiple Myeloma response rates | at 3 months
  at 3 months post-transplant according to standard response criteria. Response rates will be evaluated based on International Myeloma Working Group Uniform Response Criteria at 3 months following ASCT.
correlation between engraftment kinetics and symptom burden | 2 years
  in patients with MM who receive high-dose melphalan and fractionated CD34+ stem cell infusions
the number of CD34+ cells/Kg present | 2 years
  at the time of infusion. The difference between the number of CD34+ cells/kg given at each stem cell infusion time point and the number of CD34+ cells/kg before cryopreservation will be calculated as both a simple difference and percentage change.
To correlate the number CD34+ cells/Kg given | 2 years
  at the time of transplant with engraftment kinetics. The difference between the number of CD34+ cells/kg given at each stem cell infusion time point and the number of CD34+ cells/kg before cryopreservation will be calculated as both a simple difference and percentage change.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm